CLINICAL TRIAL: NCT05039476
Title: Study to Identify if Chemist Confessions Retinol Cream Works to Improve the Appearance of Early Signs of Aging.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chemist Confessions, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 20218Chemist
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Wrinkle; Aging

STUDY DESIGN:
Intervention Model Description: Split face intervention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retinol face cream (Active Comparator): Retinol face cream on one half of the participant's face
  Interventions: Dietary Supplement: Retinol face cream
- Placebo face cream (Placebo Comparator): Placebo face cream on one half of the participant's face
  Interventions: Dietary Supplement: Placebo face cream

INTERVENTIONS:
Dietary Supplement: Retinol face cream — Retinol face cream
  Arms: Retinol face cream
Dietary Supplement: Placebo face cream — Placebo face cream
  Arms: Placebo face cream

SUMMARY:
Chemist Confessions has developed a retinol cream with the aim to improve the appearance of early signs of aging, such as fine lines, dark spots, hyperpigmentation, and crow's feet. In this phase, Chemist Confessions plans to collect self-reported outcomes and photographic images to understand the assessment of the efficacy of treatment from the participant's perspective, and if participants see an improvement in their fine lines, wrinkles, dark spots, hyperpigmentation, and crow's feet.

DETAILED DESCRIPTION:
Based on a review of existing literature and previous studies, retinol has been found to have positive effects, however, due to study limitations, there are also conflicting results. Therefore, in this study, participants will receive Chemist Confessions retinol cream to understand if the Chemist Confessions cream has an impact on the participant's skin, and even potentially reduces fine lines, wrinkles, dark spots, hyperpigmentation, and crow's feet of the skin, and also to understand concepts considered essential by individuals taking retinol products.

ELIGIBILITY:
Inclusion Criteria:

* Female between 30-50 years old
* Must be in good general health
* Must experience early-stage wrinkles that are not treated by topical or oral prescription drugs/medication
* May experience hyperpigmentation, dark spots and dark circles
* Must maintain the following skincare routine containing: cleansing, allowed moisturizer and study specific sunscreen
* Must use study provided sunscreen daily
* Must discontinue the use of other retinoids 4 weeks before the study start date
* Must have some general knowledge of retinoid use
* Must be willing to comply with the requirements of the protocol
* Must be able to communicate in English
* Must be able to tell left from right
* Must willing to add the retinoid cream to their skincare routine
* Must provide written informed consent form (ICF)
* Is willing and able to share feedback and take skin pictures via the used technology portal
* Must be willing to refrain from using products with chemical exfoliants glycolic acid and lactic acid during the duration of the study

Exclusion Criteria:

* Unwilling to provide consent
* Unwilling to add the retinoid cream to their normal skincare routine
* Unwilling to follow the routine of the protocol
* Uses moisturizers that include chemical exfoliating ingredients such as glycolic acid, lactic acid or salicylic acid
* Use of other oral retinoids
* Use of prescription medication relevant to the skin
* Undergoing any cosmetic procedures during the study including Botox, laser or chemical peel treatments
* Deep-set of wrinkles
* Use of prescription drug (topical or oral) that is targeted at any sort of skin condition (for example retinoids)
* Is pregnant or nursing, or attempting a pregnancy
* Used retinoids before with an adverse reaction
* Has a self-identified sensitive skin type
* Has any learning and/or cognitive difficulties that prevent him/her reading and understanding questionnaires and surveys (e.g. dementia)

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female between 30-50 years old
Enrollment: 35 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Improvement of skin appearance of early signs of aging | 12 weeks
  The primary objective of this study is to understand if Chemist Confessions retinol cream is capable of improving the appearance of early signs of aging such as fine lines, dark spots, wrinkles, hyperpigmentation and crow's feet, and to determine if it helps to improve the overall skin health by promoting hydrated, brightened skin for study participants.
  To evaluate the improvement of this outcome measure VISIA imaging will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, MSc, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No